CLINICAL TRIAL: NCT00003703
Title: Phase I and Pharmacokinetics Study of SarCNU in Patients With Advanced Cancers
Brief Title: Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066810; JGH-CR97097; CR-97-0917; CR9809NI; NCI-T98-0015
Record Dates: First submitted 1999-11-01; First posted 2004-03-15 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2002-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — 2-((((2-chloroethyl)nitrosoamino)carbonyl)amino)propanamide

INTERVENTIONS:
Drug: SarCNU

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of chemotherapy using sarCNU in patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of SarCNU in patients with advanced solid malignancies. II. Determine the toxic effects of SarCNU in these patients. III. Characterize the pharmacokinetic profile of this regimen in these patients. IV. Determine any evidence of antineoplastic activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study. Patients receive oral SarCNU on days 1, 5, and 9. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of SarCNU until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at the MTD.

PROJECTED ACCRUAL: Approximately 12-36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced solid malignancy for which no curative or life-extending therapy exists No prior or concurrent CNS metastases Primary CNS tumors allowed if on a stable dose of steroids at least 2 weeks before study entry No myelodysplastic syndrome

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: More than 12 weeks Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 120,000/mm3 Hemoglobin greater than 8 g/dL Hepatic: Bilirubin normal AST and ALT less than 2.5 times upper limit of normal Renal: Creatinine less then 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: No uncontrolled cardiac disease No uncontrolled hypertension Pulmonary: DLCO and vital capacity greater than 80% predicted Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception HIV negative Oral intake at least 1,200 calories per day No recent weight loss of more than 10% actual body weight No serious concurrent illness No uncontrolled infection

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy No concurrent immunotherapy No concurrent immunomodulating agents Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) No other concurrent cytostatic or cytotoxic chemotherapy Endocrine therapy: See Disease Characteristics No concurrent hormonal therapy No concurrent dexamethasone Radiotherapy: At least 3 weeks since prior radiotherapy No prior radiotherapy to more than 25% of bone marrow No concurrent radiotherapy Surgery: At least 3 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-01; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C. Panasci, MD, Study Chair — Jewish General Hospital
Locations (1):
- Jewish General Hospital - Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Result] Panasci L, Stinson SF, Melnychuk D, Sandor V, Miller WH Jr, Batist G, Patenaude F, Bangash N, Panarello L, Alaoui-Jamali M, Sausville E. SarCNU, a nitrosourea analog on a day 1, 5, and 9 oral schedule: a phase I and pharmacokinetic study in patients with advanced solid tumors. J Clin Oncol. 2003 Jan 15;21(2):232-40. doi: 10.1200/JCO.2003.03.047. PMID 12525514